CLINICAL TRIAL: NCT06472921
Title: Effect of Early Initiation of Butylphthalide on Neural Function in Patients With Acute Ischemic Stroke -A Prospective, Multicenter, Randomized, Open-label, Blinded End Trial
Brief Title: Efficacy and Safety of Early Initiation of Butylphthalide Treatment in Patients With Acute Ischemic Stroke.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202405104
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Eligible participants with acute ischemic stroke will be randomly assigned in a 1:1 ratio to two groups: an early initiation group and a late initiation group.
  Early initiation group: Treatment with Butylphthalide Sodium Chloride Injection begins within 3 hours, administered at 100ml per dose, infused twice daily for a continuous period of 10-14 days.
  Late initiation group: Treatment with Butylphthalide Sodium Chloride Injection begins between 3-6 hours, also administered at 100ml per dose, infused twice daily for a continuous period of 10-14 days.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early initiation group (Experimental): Treatment with Butylphthalide Sodium Chloride Injection begins within 3 hours, administered at 100ml per dose, infused twice daily for a continuous period of 10-14 days.
  Interventions: Behavioral: Butylphthalide treatment initiation time
- Treatment with Butylphthalide Sodium Chloride Injection begins within 3 hours, administered at 100ml (Other): Treatment with Butylphthalide Sodium Chloride Injection begins within 3 hours, administered at 100ml per dose, infused twice daily for a continuous period of 10-14 days.
  Interventions: Behavioral: Butylphthalide treatment initiation time

INTERVENTIONS:
Behavioral: Butylphthalide treatment initiation time — Eligible participants with acute ischemic stroke will be randomly assigned in a 1:1 ratio to two groups: an early initiation group (<3 hours) and a late initiation group (3-6 hours).

SUMMARY:
This study is a prospective, multicenter, randomized, open-label, blinded-endpoint trial designed to evaluate the difference in efficacy of Butylphthalide Sodium Chloride Injection treatment initiated early (<3 hours) versus late (3-6 hours) in patients with acute ischemic stroke. The aim is to determine the optimal timing window for neuroprotective therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, gender not specified;
2. Clinically diagnosed with acute ischemic stroke;
3. Stroke onset within 3 hours;
4. NIHSS score at enrollment between 4-25 points, with Item Ia ≤1 point;
5. Pre-stroke mRS score ≤1 point;
6. Participants and their representatives capable and willing to sign an informed consent form.

Exclusion Criteria:

1. Confirmed intracranial hemorrhage within the past 3 months, including intracerebral hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, and subdural/epidural hematoma;
2. Known severe hepatic or renal dysfunction or individuals undergoing dialysis for various reasons (severe hepatic dysfunction defined as ALT levels >3 times the upper limit of normal or AST levels >3 times the upper limit of normal; severe renal dysfunction defined as serum creatinine >3.0 mg/dl [265.2 μmol/L] or glomerular filtration rate [GFR] <30 ml/min/1.73m²);
3. Systolic blood pressure <90 mmHg or >220 mmHg;
4. Presence of bradycardia (heart rate below 60 beats per minute) or sick sinus syndrome;
5. History of drug or food allergies, including known allergies to the components of the study medication;
6. Treatment with medications containing Butylphthalide following the onset of the current stroke episode;
7. Congenital or acquired hemorrhagic disorders, coagulation factor deficiencies, thrombocytopenia, or similar conditions;
8. Pregnant or breastfeeding individuals, or those planning to become pregnant within the next 90 days;
9. Severe psychiatric disorders or dementia that preclude understanding of informed consent or compliance with follow-up procedures;
10. Concurrent malignancy or severe systemic disease with a life expectancy of less than 90 days;
11. Participation in another interventional clinical study within the last 30 days before randomization, or currently participating in another interventional clinical study;
12. Any other reason deemed by the investigator as unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with an mRS score of 0-2 | 90±7 days post-randomization

SECONDARY OUTCOMES:
Proportion of participants with an mRS score of 0-1 | 90±7 days post-randomization
Changes in NIHSS scores | at 6±1 days and 12±2 days compared to baseline
Proportion of participants with an improvement of ≥4 points in NIHSS scores | at 6±1 days and 12±2 days
Early neurological deterioration | at 24±2 hours and 6±1 days post-randomization
Proportion of participants with ineffective recanalization | at 90±7 days post-randomization
Proportion of participants with recurrent ischemic stroke | at 90±7 days post-randomization
Proportion of combined vascular events (recurrent stroke, myocardial infarction, and vascular death) | at 90±7 days post-randomization
Difference in cerebral infarction volume size | between baseline and 12±2 days post-randomization
Quality of life (EQ-5D) scores | at 90±7 days post-randomization

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha